CLINICAL TRIAL: NCT05250869
Title: Comparative Quantification of MTX and Its Metabolites in Acidified vs. Non-acidified Blood Samples Post Glucarpidase Using HPLC/MS
Brief Title: Comparative Quantification of MTX and Its Metabolites Post Glucarpidase
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Stefan Schwartz, PD Dr. Stefan Schwartz, Charite University, Berlin, Germany
Other Study IDs: EA4/258/21
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Lymphoma; Acute Lymphatic Leukemia
Keywords: Preanalytical Conditions
MeSH Terms: conditions — Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HPLC/MS — Quantification of MTX and its metabolites by HPLC/MS under various preanalytical conditions

SUMMARY:
Acidification (i.e., addition of hydrochloric acid) of plasma samples from patients who have received Glucarpidase post high-dose MTX treatment is regarded as a necessary preanalytic step to avoid further in vitro enzymatic cleavage of MTX. However, it is unclear whether this acidification step is essential. A comparative study, which evaluates concentrations of MTX and its metabolites in paired (acidified versus non-acidified) plasma samples, has not yet been performed. Processing plasma samples without acidification would facilitate quantification of MTX, including plasma samples from patients treated at centers without adequate laboratory facilities.

DETAILED DESCRIPTION:
Stored plasma samples (paired - acidified and non-acidified) from the specimens collection ('Tumorbiobank') of the Charité Comprehensive Cancer Center will be analysed by HPLC/MS.

A total of 136 samples from patients post Voraxaze across 3 levels of MTX concentrations:

30 without additive, 10 with 0.9% NaCl, 30 with HCl (stored at -80C) 9 without additive, 9 with HCl (stored at +4C and analysed after 3-5 days) 9 without additive, 9 with HCl (stored at -20C and analysed after 3-5 days) 30 with HCl (stored at +4C versus ambient temperature)

ELIGIBILITY:
Inclusion Criteria:

* Treatment with Glucarpidase

Exclusion Criteria:

* Lacking patient consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with high-dose Methotrexate and Glucarpidase
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Consistency of MTX concentrations in paired acidified vs. non-acidified samples | within 3 days of Glucarpidase treatment
  Comparison of MTX/metabolite concentrations

SECONDARY OUTCOMES:
Consistency of MTX concentrations in paired samples stored at -80C vs. +4C vs. ambient temperature | within 3 days of Glucarpidase treatment
  Comparison of MTX/metabolite concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Result] Knornschild FL, Liebig S, Kiessling P, Prpic M, Kim T, Keller U, Kappert K, Schwartz S, Jahic A. Simplified preanalytical laboratory procedures for therapeutic drug monitoring (TDM) in patients treated with high-dose methotrexate (HD-MTX) and glucarpidase. Clin Chem Lab Med. 2024 Jul 15;63(1):e11-e15. doi: 10.1515/cclm-2024-0523. Print 2025 Jan 29. No abstract available. PMID 38997789